CLINICAL TRIAL: NCT01042119
Title: Short- and Longterm Results After Intravesical Injection of Botulinum Neurotoxin Type A for Treating Therapy Refractory Overactive Bladder in Females - a Retrospective Study
Brief Title: Intravesical Injection of Botox for Treating Therapy Refractory Overactive Bladder in Females
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Scheiner, David, Dr. med., University Hospital of Zurich, Clinic for Gynaecology
Other Study IDs: FHKUSZ15-2009
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Overactive Bladder Syndrome
Keywords: botulinum neurotoxin type A; BoNT/A; Botox; overactive bladder syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Botox: patients who received intravesical injections of botulinum neurotoxin type A

SUMMARY:
The neurotoxin Botox (botulinum neurotoxin type A) is shown to be effective in the treatment of therapy refractory overactive bladder syndrome. Our data suggests a longer during efficacy than known from the use in striated muscle.

The aim of our study is to analyze short- and longterm efficacy after Botox treatment and to evaluate risk factors for non-responders and side effects such as urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* intravesical treatment with Botox at our clinic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who received at our clinic treatment with intravesical injection of Botox for idiopathic overactive bladder syndrome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
duration of effect of Botox | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David A Scheiner, MD, Principal Investigator — University Hospital of Zurich, Clinic for Gynaecology
Locations (1):
- University Hospital of Zurich, Clinic for Gynaecology, Zurich, Switzerland